CLINICAL TRIAL: NCT01829620
Title: Military Continuity Project (MCP): A Suicide Prevention Study
Brief Title: Military Continuity Project
Acronym: MCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Military Suicide Research Consortium (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kate Comtois, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001901; W81XWH1020181/089009520027450 (Other Grant/Funding Number: Department of Defense/Florida State University)
Record Dates: First submitted 2013-03-30; First posted 2013-04-11 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Suicidal Ideation Active; Suicidal and Self-injurious Behavior
Keywords: suicide; suicide intervention; suicide prevention; military; military suicide; caring letters; caring contacts; text messages
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Suicide Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): The Treatment as Usual (TAU) control group will reflect current clinical practices for treating suicidal Soldiers and Marines.
  Interventions: Behavioral: TAU
- Continuing Contacts via Text (CCVT)+TAU (Experimental): The intervention group will receive Continuing Contacts via Text (CCVT) in addition to Treatment as Usual (TAU).
  Interventions: Behavioral: CCVT+TAU

INTERVENTIONS:
Behavioral: TAU — This is standard outpatient mental health care that is routinely provided in study site outpatient clinics.
  Arms: Treatment as Usual (TAU)
Behavioral: CCVT+TAU — Participants in the CCVT + TAU condition will receive caring texts at 1 day, 1 week, 1, 2, 3, 4, 6, 8, 10, & 12 months, and on their birthday. Text messages will indicate a general concern for the individual and a link to a website with general resources including behavioral health and crisis services.
  Participants in both conditions will continue to receive usual behavioral health care according to standard operating procedures.
  Arms: Continuing Contacts via Text (CCVT)+TAU

SUMMARY:
The investigators propose to utilize text messaging to create and investigate the efficacy of a Continuing Contacts via Text (CCVT) intervention that extends the continuity of care for Service Members with a recent suicide attempt and/or reported suicidal ideation by sending them non-demanding caring text messages at regular intervals over a 12-month period. Participants will be randomly assigned to receive Continuing Contacts via Text (CCVT) in addition to Treatment as Usual (TAU) or TAU alone.

Aim 1: To determine if the addition of 12 months of CCVT to TAU (CCVT+TAU) results in lower rates of suicidal ideation and behavior relative to TAU alone.

* Hypothesis 1a: Participants assigned to CCVT+TAU compared to TAU alone will experience reduced suicidal ideation at 12-month follow-up.
* Hypothesis 1b: Over the 12 months following study enrollment, a smaller proportion of participants assigned to CCVT+TAU vs. TAU alone will have suicide risk incidents (i.e., those requiring medical evacuation or hospital admission).
* Hypothesis 1c: Over the 12 months following study enrollment, CCVT+TAU vs. TAU alone will have fewer total number of suicide risk incidents requiring medical evacuation or hospital admission.

Aim 2: To test two proposed mechanisms of action of CCVT outcome: 1) reduced "thwarted belongingness" and 2) increased engagement in behavioral health services.

* Hypothesis 2a: The effect of CCVT+TAU compared to TAU alone will be mediated by reductions in "thwarted belongingness" from pre to post-study.
* Hypothesis 2b: The effect of CCVT+TAU compared to TAU alone will be mediated by increased use of outpatient behavioral health services in the CCVT+TAU condition.

DETAILED DESCRIPTION:
Apparent increases in suicide attempts and death by suicide among active duty Service Members have gained considerable attention from the media, members of Congress, and the Department of Defense. Identifying and intervening with individuals thinking of suicide (as well as those engaging in suicidal behavior) is key to preventing suicide in Service Members. Intervention through caring contacts (e.g., letters, phone calls) have efficacy showing they may be an important adjunct or alternative to outpatient care. Caring contact interventions have been shown in previous studies to decrease suicidal ideation and attempts and initial pilot data have shown positive results in military populations.

Text messaging, a low-cost means of sending brief messages (160 characters) to any owner of a mobile phone, has been investigated as an intervention for improving attendance to medical appointments and adherence to treatment in medical populations. As our current military population is a young, mobile, and increasingly technologically savvy population, and with the growing support behind text messaging as a feasible and effective mode of behavioral intervention, the pairing of text messaging and caring contact interventions warrants further research.

The investigators plan to randomize 800 participating Service Members to one of the two treatment conditions (i.e., CCVT+TAU or TAU alone) to test the efficacy of this intervention. Measured endpoints will include suicide risk incident requiring medical evacuation or hospitalization, suicidal ideation as identified by the follow-up assessment battery, "thwarted belongingness" as identified by The Interpersonal Needs Questionnaire, outpatient behavioral health care utilization, and death.

ELIGIBILITY:
INCLUSION CRITERIA:

* Active duty, Reserve, National Guard
* 18 or more years of age
* Identification to a behavioral health, counseling, or medical service (inpatient, outpatient, or emergency) with suicidal ideation or a suicide attempt
* Has current suicidal ideation as defined by the Scale for Suicidal Ideation-Current (SSI-C)
* Has mobile phone or pager where he or she can receive 11 text messages in a year free of cost or at a fee he or she does not consider burdensome

EXCLUSION CRITERIA:

* Does not speak and read English well enough to consent and to understand texts in English
* Too cognitively impaired at best mental status during treatment to consent to participate (i.e., brain damage, psychosis, dementia, or other cause)
* Treating clinician evaluates the intervention as contra-indicated (e.g., paranoia exacerbated by being contacted)
* Prisoner or otherwise under judicial order where study participation could not be considered to be truly voluntary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Scale for Suicide Ideation - Current (SSI-C) | 12 months
  The SSI-C is an interviewer-administered scale that measures a Service Member's suicidal ideation at its worst point in the past 2 weeks.
Treatment History Interview (THI) | 12 months
  The THI captures the subject's treatment history. The investigators have modified a version to more appropriately capture the services Service Members are likely to receive, the Treatment History Interview - Military (THI-M). Primary outcome measured by the THI-M is suicide risk incidents (inpatient admission or medical evacuation to prevent suicide)

SECONDARY OUTCOMES:
Suicide Attempt Self-Injury Count (SASI-Count) | 12 months
  The SASI-Count is an interviewer-administered brief instrument that creates a thumbnail sketch of a participant's history of self-directed violence (SDV) by assessing the first, most recent, and most severe acts of SDV during a specified time period, including the date, method, and suicidal intent of the act. This is followed by an assessment of SDV across 12 methods (e.g., cutting, hanging or strangling, firearm), generating counts by method and then classifying each act by suicidal intent (no, ambivalent, or clear intent). Across each method, the most lethal event is coded on a 1-6 scale in which "1" is "very low" (e.g., head banging) and "6" is "severe" (e.g., pulling the trigger of a loaded gun aimed at a vital area). A "Lifetime" version of the instrument was used at baseline, assessing all lifetime acts of SDV. A "Recent" version assessed SDV in the past year at baseline and at 12-month follow-up.
Scale for Suicide Ideation - Worst (SSI-W) | 12 months
  The SSI-W focused on worst-point ideation lifetime when administered at enrollment. At 12 months, the SSI-W captured worst-point ideation, if any, between baseline and follow-up. The SSI-W was added as an outcome after the first 35 cases completed follow-up upon learning it was becoming a standard in clinical trials using the SSI.
Interpersonal Needs Questionnaire (INQ) | 12 months
  The INQ, developed by Joiner and colleagues, will be used to measure beliefs about the extent to which individuals feel connected to others and feel like a burden on the people in their lives. Change in thwarted belongingness is being tested as a mediator of outcome.
Treatment History Interview (THI) | 12 months
  The THI captures the subject's treatment history. The investigators have modified a version to more appropriately capture the services Service Members are likely to receive, the Treatment History Interview - Military (THI-M). Secondary outcomes measured by the THI-M include outpatient behavioral health treatments received by participants and emergency department visits.
Client Satisfaction Questionnaire (CSQ) | 12 months
  The CSQ is a brief eight-item questionnaire, which is used frequently for evaluating standard community mental health care. The CSQ will help determine if the caring texts improve treatment satisfaction.

OTHER OUTCOMES:
Demographic Data Schedule (DDS) | Baseline
  The DDS obtains a wide range of demographic data.
Mobile Phone Use Questionnaire | 12 months
  A series of questions characterizing the Service Member's mobile and texting capacity and history will be included to determine that they are likely to receive the study texts and contextualize the receipt of these texts in terms of their frequency of text, phone, and other technology use.
Military Suicide Research Consortium Common Data Elements (MRSC CDE) | 12 months
  The MRSC CDE includes items regarding suicidal behavior, behavioral health and traumatic brain injury symptoms, and hopelessness that are to be included in all MRSC-funded studies.
Text Message Reception Survey | 12 months
  The Text Message Reception Survey is a short questionnaire regarding whether or not the participant received text messages from the study staff, and attitudes about the text messages.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Anne Comtois, PhD, MPH, Principal Investigator — University of Washington; Richard K Ries, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Marine Corps Air Ground Combat Center Twentynine Palms, Twentynine Palms, California
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Marine Corps Base Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina

REFERENCES:
- [Background] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Background] Motto JA. Suicide prevention for high-risk persons who refuse treatment. Suicide Life Threat Behav. 1976 Winter;6(4):223-30. PMID 1023455
- [Background] Luxton DD, Kinn JT, June JD, Pierre LW, Reger MA, Gahm GA. Caring Letters Project: a military suicide-prevention pilot program. Crisis. 2012 Jan 1;33(1):5-12. doi: 10.1027/0227-5910/a000093. PMID 21940244
- [Derived] Comtois KA, Kerbrat AH, DeCou CR, Atkins DC, Majeres JJ, Baker JC, Ries RK. Effect of Augmenting Standard Care for Military Personnel With Brief Caring Text Messages for Suicide Prevention: A Randomized Clinical Trial. JAMA Psychiatry. 2019 May 1;76(5):474-483. doi: 10.1001/jamapsychiatry.2018.4530. PMID 30758491